CLINICAL TRIAL: NCT00199667
Title: APOMYGRE : Multicenter, Randomized, Open-Label Study of MMF Therapeutic Follow-up's Interest in the the 12 First Months in Kidney Transplantation
Brief Title: Concentration Controlled Versus Fixed Dose of MMF in Kidney Transplant Recipients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Limoges (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I02013
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Kidney Transplant Recipients
Keywords: MMF, Monitoring, area under curve (AUC), kidney transplantation
MeSH Terms: interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: Mycophenolate Mofetil

SUMMARY:
Acumulating data suggest that thrapeutic drug therapeutic may optimize efficacity and tolerance of MMF. It could guarantee better exposure to the drug in the first 3 months and then minimize side effects in the long term. However definitive proof is still lacking. We conducted a randomized study in 11 french centers and included 137 kidney transplant recipients (PRA<50%) receiving a classical immunosuppressant regimen with basiliximab, Csa, MMF and steroids. The "fixed dose" group received 2 g of MMF a day. The "concentration controlled" group received MMF dose adapted to the area under the concentration curve (AUC) of MPA, with a target of 40 h.mg/L. After transplantation AUCs were calculated with a Bayesian estimator using a 3-point limited sampling strategy on day 7, 14, and months 1, 3, 6 , 12 in both groups (values note communicated to the physicians in the "fixed dose" group.

ELIGIBILITY:
Inclusion Criteria:

* patients received a first or a second kidney transplantation
* patients with panel reactive antibody <or= 50 %
* patients with cellcept treatment since fewer 3 days
* patients receiving or being received ciclosporine treatment
* patients without retention, important hepatic cytolysis
* patients without post-surgical complication or intercurrent disease
* informed consent signed

Exclusion Criteria:

* patients included in other study
* patients with MMF or mycophenolic acid hypersensibility or MMF contraindication
* patients with gastroduodenal disorder before the beginning of the study
* pregnant women or without contraception
* patients with rapamycin or analogous
* patients with toxicomania or psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137
Dates: Start 2002-10

PRIMARY OUTCOMES:
immunosuppressant treatment fealure (kidney rejection, adverse events, death, graft lost).

SECONDARY OUTCOMES:
renal fonction evolution

CONTACTS AND LOCATIONS:
Overall Officials: Yann LE MEUR, MD, Principal Investigator — University Hospital, Limoges
Locations (11):
- France (11):
  - Néphrologie, Amiens
  - Néphrologie, Angers
  - Néphrologie, Caen
  - Néphrologie, Limoges
  - Néphrologie, Paris
  - Néphrologie, Poitiers
  - Néphrologie, Reims
  - Néphrologie, Rouen
  - Néphrologie, Strasbourg
  - Néphrologie, Toulouse
  - Néphrologie, Tours